CLINICAL TRIAL: NCT03033238
Title: Multicenter Osteoarthritis Study (MOST) Second Renewal
Brief Title: Multicenter Bone and Joint Health Study
Acronym: MOST
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Iowa (Other); University of Alabama at Birmingham (Other); Boston University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: U01AG019069 (NIH); U01AG019069 (NIH)
Record Dates: First submitted 2016-12-01; First posted 2017-01-26 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis,Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Existing Cohort biospecimens were collected at enrollment, 30-month and 60-month follow-up. New Cohort biospecimens will be collected at 144-month which will be their enrollment visit).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Early or mild knee symptoms: Existing Cohort study participants (3,026) were enrolled in 2003-2005, Surviving participants without endstage knee osteoarthritis will be asked to participate in the 144-, 152-, 160- and 168-month follow-up contacts [2,660 were enrolled].
  New Cohort study participants (1,500) will be recruited and enrolled in 2016-2018 [1,525 were enrolled].

SUMMARY:
The purpose of this study is to investigate opportunities for prevention and treatment of knee osteoarthritis (OA) by evaluating potentially modifiable risk factors for disease and poor pain and physical function outcomes especially among those with early or mild knee symptoms. The goal of the study is to find novel strategies to prevent disease at an early stage and to limit the impact of disease once it has occurred.

DETAILED DESCRIPTION:
MOST study participants in the "Existing Cohort" (3,026 subjects) were enrolled in the original study in 2003-2005. Surviving Existing Cohort participants without end-stage knee osteoarthritis will be asked to participate in the 144-, 152-, 160- and 168-month follow-up contacts. In addition, in 2016-2018 the cohort will be enriched by the recruitment of an additional 1,500 "New Cohort" participants with early or mild knee symptoms. The goal of the study is to find novel strategies to prevent disease at an early stage.

ELIGIBILITY:
Inclusion Criteria for "New Cohort" Participants:

* Age 45 to 69 Years (Adult, Senior)
* Males and Females
* Healthy Volunteers
* Community-based Sample

Exclusion Criteria for "New Cohort" Participants:

* Rheumatoid or inflammatory arthritis (based on self-report and use of medications specific to these conditions)
* Serious health condition e.g., end-stage renal disease, etc. that would likely limit follow-up to less than 2-3 years
* Plan to relocate out of geographic region in next 3 years
* Not able to walk without the aid of a person or assistive device
* Knee joint replacement surgery in either knee
* Neither knee fits in the MRI knee coil (determined during Screening Visit).
* Not competent to give informed consent
* Advanced structural tibiofemoral or patellofemoral knee OA disease (KL grade 3 or 4) in either knee (Determined by Knee X-ray Screening)

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The purpose of this study is to investigate opportunities for prevention and treatment of knee osteoarthritis by evaluating potentially modifiable risk factors for disease and poor pain and physical function outcomes especially among those with early or mild knee symptoms. The goal of the study is to find novel strategies to prevent disease at an early stage and to limit the impact of disease once it has occurred.
Sampling Method: Probability Sample
Enrollment: 4185 (Actual)
Dates: Start 2003-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Worsening knee pain | Change from baseline (144-month) at ≥2 follow-up contacts (152-, 160-, 168-month follow-up contacts)
  Worsening knee pain defined as reaching minimally clinically important difference (MCID) for worsening on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain questionnaire
Incident cartilage loss on MRI | Change from baseline (144-month) at 168-month follow-up contact
  Incidence of cartilage loss on MRI extending to the bone
Function loss | Change from baseline (144-month) at ≥2 follow-up contacts (152-, 160-, 168-month follow-up contacts)
  Defined as minimally clinically important difference (MCID) for worsening on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function questionnaire

SECONDARY OUTCOMES:
Onset of constant knee pain | Change from baseline (144-month) at ≥2 follow-up contacts (152-, 160-, 168-month follow-up contacts)
  Self- report
Worsening on MRI | Change from baseline (144-month) at 168-month follow-up contact
  Worsening cartilage scores, bone marrow lesion, or meniscal damage
Worsening on X-ray | Change from baseline (144-month) at 168-month follow-up contact
  Increased Kellgren-Lawrence (KL) grade score, new KL grade 2 score, or semi-quantitative joint space loss in any compartment
New onset knee buckling | Change from baseline (144-month) at ≥1 follow-up contact (152-, 160-, 168-month follow-up contacts)
  Self-report
New repeated falls | Change from baseline (144-month) at ≥1 follow-up contact (152-, 160-, 168-month follow-up contacts)
  Self-report

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nevitt, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Iowa, Iowa City, Iowa
  - Boston University School of Medicine, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Anonymized clinical data will be shared via The NIA Biobank (https://agingresearchbiobank.nia.nih.gov/). MOST Existing Cohort data from previous grant cycles will be available in mid 2021. For more information visit MOST Online (https://most.ucsf.edu).
Supporting Information: Study Protocol
Access Criteria: See NIA Biobank website
URL: https://agingresearchbiobank.nia.nih.gov/

REFERENCES:
- [Derived] Rabe KG, Stockman TJ, Kern AM, Wirth W, Eckstein F, Sharma L, Lynch JA, Nevitt MC, Anderson DD, Segal NA. Longitudinal Relationship Between Tibiofemoral Contact Stress at Baseline and Worsening of Knee Pain Over 84 Months in the Multicenter Osteoarthritis Study. Am J Phys Med Rehabil. 2022 Aug 1;101(8):726-732. doi: 10.1097/PHM.0000000000001899. Epub 2021 Oct 8. PMID 34620738